CLINICAL TRIAL: NCT04509817
Title: Efficacy and Safety of Acupuncture on Oligomenorrhea Due to Polycystic Ovary Syndrome: an International Multicenter, Pilot Randomized Controlled Trial
Brief Title: Acupuncture for Oligomenorrhea Due to Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government); Dongzhimen Hospital, Beijing (Other); Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Chunlan Jin, Associated professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GH201802; KHNMCOH 2017-12-003 (Other: Kyung Hee University Hospital at Gangdong)
Record Dates: First submitted 2020-07-01; First posted 2020-08-12 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Polycystic Ovary Syndrome; Oligomenorrhea
Keywords: Polycystic ovary syndrome; Oligomenorrhea; Acupuncture
MeSH Terms: conditions — Polycystic Ovary Syndrome; Oligomenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture+Usual care (Experimental): Subjects in experimental group will receive a standardized acupuncture treatment, 10 times per 4 weeks for 16 weeks with a total of 40 sessions in addition to usual care.
  Interventions: Device: Acupuncture+Usual care
- Usual care (Active Comparator): Subjects in control group will receive usual care only.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Device: Acupuncture+Usual care — Acupuncture intervention Disposable, sterilized needles (0.25×40 mm and 0.30×50 mm) will be used and selected acupoints will include GV20, CV4, and bilateral BL32, ST25, ST29, EX-CA1, LI4, LR3, SP6, SP9. Subject will be prone position first and BL32 will be inserted with an angle of 30-45° in an inferomedial direction and a depth of 30-50 mm. Once the subject has a needle sensation ('De-qi'), the needle will be removed immediately. Then the subject will be supine position, and GV20, CV4, ST25, ST29, EX-CA1, LI4, LR3, SP6, SP9 will be needled with a depth of 10-40mm. After subject feel 'De-qi', the needles will be placed for 20 min to maintain the stimulation.
  Usual care intervention The subjects will receive the health advice including diet with regular meal, enough sleep, and appropriate exercise.
  Behavioral: Usual care Usual care intervention The subjects will receive the health advice including diet with regular meal, enough sleep, and appropriate exercise.
  Arms: Acupuncture+Usual care
Behavioral: Usual care — Usual care intervention The subjects will receive the health advice
  Arms: Usual care

SUMMARY:
This study is an international multicenter, pilot randomized, assessor-blind, controlled trial, which is aimed to preliminarily investigate the efficacy and safety of acupuncture on oligomenorrhea due to polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
A total of 60 subjects will be recruited and randomly allocated into experimental or control group with 30 subjects respectively. The subjects in experimental group will receive a standardized acupuncture treatment plus usual care, whereas the ones in control group will be managed only with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Oligomenorrhea (menstrual cycle> 35 days or less than 8 cycles per year) plus at least one of the following two criteria; hyperandrogenism (clinical, biochemical, or both) and/or polycystic ovarian morphologic features [12 or more antral follicles (2 to 9 mm in diameter) in either ovary, an ovarian volume that is greater than 10 ml in either ovary, or both]
* 20-40 years of age
* Voluntary agreement to participate in this trial

Exclusion Criteria:

* Pregnancy, labor or breastfeeding within the past 3 months
* Intake of oral contraceptive or ovulation inducing agent within the past 3 months
* Severe oligomenorrhea with menstrual period over 3 months
* Menstruation during more than 8 days
* Premature ovarian failure
* Resistant thyroid disease, Cushing's disease, congenital adrenal hyperplasia, or hyperprolactinemia
* Ovarian tumor or adrenal tumor that cause hyperandrogenemia
* Hemorrhagic disease
* Severe cardiac, pulmonary, hepatic, or renal diseases, central nervous system disorders, or intake of psychoactive drug
* Acupuncture treatment within the past one month
* Participation in other clinical trial within the past 3 months
* Other conditions judged to be inappropriate for the clinical study by the investigators

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Menstrual Frequency (cycles/month) | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Menstrual cycle improvement will be assessed by menstrual frequency (cycle/month).

SECONDARY OUTCOMES:
Change in Menstrual Period | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Menstrual period is assessed in days from the 1st day of menstruation cycle to 1st day of the next menstruation cycle.
Change in Estradiol (E2) | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Change in the level of serum estradiol in pg/mL
Change in Luteinizing Hormone (LH) | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Change in the level of serum luteinizing hormone (LH) in mIU/mL
Change in Serum Follicle Stimulating Hormone (FSH) | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Change in the level of serum follicle stimulating hormone (FSH) in mIU/mL
Change in Free Testosterone (T) | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Change in the level of serum free testosterone (T) in ng/mL
Change in LH/FSH Ratio | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  The ratio is calculated based on the value of LH and FSH.
Change in Antral Follicle Count (AFC) in the Ovary and Ovarian Volume | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Change in the number of antral follicles of the ovary and ovarian volume by ultrasound imaging.
Change in Body mass index (BMI) | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Body Mass Index (BMI) is defined as the body weight divided by the square of height, and expressed in kg/m2.
Change in Waist Hip Ratio (WHR) | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  The ratio is calculated based on the length of waist and hip.
Change in acne severity evaluated by Pillsbury acne grading system | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Acne severity is assessed by Pillsbury acne grading system. The grade of Pillsbury acne grading system ranges from 0 to 4. The high-scored grade means the more severe acne (i.e., grade 0 is considered to be normal, and grade 4 is considered severe).
Change in quality of life evaluated by the 36-Item Short Form Health Survey (SF-36) | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  SF-36 is a 36-item, patient-reported survey of patient health, which consists of eight sections. The score of SF36 ranges from 0 to 100. The higher the score, the less disability, i.e., a score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Adverse events | up to 32 weeks
  All expected or unexpected adverse events in both groups will be measured at every study visit.
  * Assessment of severity: mild, moderate, severe
  * Assessment of relation: definitely related, probably related, possibly related, probably not related, definitely not related, unknown.
Incidence of abnormal complete blood count | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  The incidence of patients with abnormal complete blood count which includes the white blood cells count in ×10^9/L, the red blood cells count in ×10^12/L, platelets count in number ×10^9/L, and hemoglobin in g/L, and hematocrit in %.
Incidence of abnormal erythrocyte sedimentation rate | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Incidence of patients with abnormal erythrocyte sedimentation rate in mm/h.
Incidence of abnormal renal function | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Incidence of abnormal lactate dehydrogenase and creatine phosphokinase. Incidence of patients with abnormal lactate dehydrogenase in U/L, and creatinine phosphokinase in U/L.
Incidence of abnormal liver function | Baseline, post-intervention (16 weeks), follow-up (32 weeks)
  Incidence of patients with abnormal liver function evaluated by serum aspartate aminotransferase in U/L, alanine aminotransferase in U/L, and γ-glutamyl-transpeptidase in U/L, alkaline phosphatase U/L, total protein in g/L, and albumin in g/L.

CONTACTS AND LOCATIONS:
Overall Officials: Chunlan Jin, MD, Principal Investigator — Institute of acupuncture and moxibustion, CACMS
Locations (3):
- China (2):
  - Dongzhimen Hospital, Beijing, Beijing Municipality
  - Institute of acupuncture and moxibustion, Beijing, Beijing Municipality
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The agreement for sharing IPD is not designed to be signed in informed consent form.

REFERENCES:
- [Derived] Park KS, Gang W, Kim PW, Yang C, Jun P, Jung SY, Kwon O, Lee JM, Lee HJ, Lee SJ, Jing X, Zhang N, Hu J, Zhao J, Pang R, Jin C, Lee JH. Efficacy and safety of acupuncture on oligomenorrhea due to polycystic ovary syndrome: An international multicenter, pilot randomized controlled trial. Medicine (Baltimore). 2022 Feb 18;101(7):e28674. doi: 10.1097/MD.0000000000028674. PMID 35363161